CLINICAL TRIAL: NCT07143474
Title: A Randomized Double-blind Placebo Controlled Clinical Study to Evaluate the Impacts of RhizomK as Compared to Placebo on Testosterone Levels, the Anabolic Response to Exercise and Overall Quality of Life in Physically Active Healthy Males
Brief Title: Effect of RhizomK on Testosterone Levels, the Anabolic Response to Exercise and Overall Quality of Life in Physically Active Healthy Males
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Dr Debasish Hota, Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: T/IM-NF/Pharm/25-26/29
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Adult Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group RhizomK (Experimental)
  Interventions: Drug: RhizomK
- Group Placebo (Placebo Comparator)
  Interventions: Other: Plcebo

INTERVENTIONS:
Drug: RhizomK — RhizomK 50 mg once daily
  Arms: Group RhizomK
Other: Plcebo — Placebo matching to RhizomK
  Arms: Group Placebo

SUMMARY:
Given that testosterone is a key modulator of muscle protein synthesis and overall anabolic response to resistance training, any natural intervention that boosts testosterone levels could logically contribute to improved exercise performance, lean muscle gain, and subjective vitality. 13 However, despite encouraging preclinical and ethnopharmacological data, clinical validation of Curculigo extract in human participants-especially in the context of exercise and lifestyle enhancement-is lacking. A novel extract of Curculigo orchioides (commercially known as RhizomK™) has been developed. This randomized, double-blind, placebo-controlled study seeks to bridge this crucial gap by evaluating the efficacy and safety of RhizomK™ supplementation in healthy, physically active males. The findings of this study have the potential to substantiate RhizomK™ as a scientifically supported dietary intervention for enhancing hormonal balance, physical performance, and well-being in men who are not candidates for pharmacological therapy but are seeking to optimize their health through lifestyle and supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Male sex, aged 21 to 40 (inclusive)
* Currently engaged in, and has been engaged in resistance training
* (i.e., weightlifting), training three or more times per week for at least
* the prior 12 months.
* Healthy subject (no medical conditions that per the PI assessment).
* No significant past medical history
* No significant past surgical history that in the opinion of the PI
* would preclude study participation.
* Passes the screening with Physical Activity Readiness questionnaire (PAR-Q)
* Not currently or recently (within the prior eight-weeks) taken a
* dietary supplement that is purported to increase testosterone
* levels.
* Agrees to follow and adhere to the study directions.
* Agrees that their study visits will be scheduled at a similar time of the day
* to minimize and potential circadian rhythm impacts.

Exclusion Criteria:

* Takes any prescribed medication or over-the-counter medication which is known to affect testosterone levels.
* Positive medical history of heart disease/cardiovascular disease, high blood pressure (140/90 or greater mmHg), kidney disease, hepatic impairment or disease, or Type I or Type II diabetes or any other medical condition or diagnosis that the PI would deem exclusionary.
* Positive medical history of unstable thyroid disease, previously diagnosed major affective disorder, psychiatric disorder that required hospitalization in the prior year, immune disorder (i.e., HIV/AIDS), a history of cancer (except localized skin cancer without metastases or in situ cervical cancer within 5 years prior to screening visit.
* Positive medical history for any gastrointestinal disease or illness Positive history of gastrointestinal surgery that is known to alter or impact the digestion, absorption of nutrients and or fluids (i.e., gastric bypass).
* History of hospitalization or in-patient or out-patient treatment for alcohol dependence or drug addiction over the past one year.
* History of hospitalization or in-patient treatment for depression or any mental health related condition within the past one year.
* Allergic to any of the ingredients in the study product.
* Subject is unwilling to follow study directions.

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study is being conducted to understand the effect of the drug on testosterone levels and anabolic response
Enrollment: 60 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Serum testosterone levels | 4 weeks
  A basal pre- intervention Saliva sample will be obtained for analysis of basal (resting) testosterone levels. One hour after ingestion of the assigned study product, the subject will undergo an acute resistance exercise routine. Resistance exercise will include the Leg Press. The post resistance-exercise session Salivary/Serum Testosterone samples within ~30 minutes of completing the exercise routine will be collected.

SECONDARY OUTCOMES:
Serum cortisol levels | 4 weeks
  A basal pre- intervention Saliva sample will be obtained for analysis of basal (resting) cortisol levels. One hour after ingestion of the assigned study product, the subject will undergo an acute resistance exercise routine. Resistance exercise will include the Leg Press. The post resistance-exercise session Cortisol samples within ~30 minutes of completing the exercise routine will be collected.
Quality of life using SF-36 (Short Form 36-Item Health Survey) | 4 weeks
  The SF-36, or 36-Item Short Form Survey, is a widely used patient-reported outcome measure (PROM) that assesses health status. It's a multi-purpose questionnaire with 36 items assessing eight health concepts: physical functioning, limitations in social activities, limitations in usual role activities, bodily pain, general mental health, vitality, and general health perceptions.
Exercise performance | 4 weeks
  1-repetition maximum (1-RM) determined for the leg press
Adverse effect | 4 weeks
  Proportion of patients in each group experiencing adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Debasish Hota, DM, Principal Investigator — AIIMS, Bhubaneswar
Locations (1):
- All India Institute of Medical Sciences, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hackney AC. Hypogonadism in Exercising Males: Dysfunction or Adaptive-Regulatory Adjustment? Front Endocrinol (Lausanne). 2020 Jan 31;11:11. doi: 10.3389/fendo.2020.00011. eCollection 2020. PMID 32082255
- [Background] Osterberg EC, Bernie AM, Ramasamy R. Risks of testosterone replacement therapy in men. Indian J Urol. 2014 Jan;30(1):2-7. doi: 10.4103/0970-1591.124197. PMID 24497673